CLINICAL TRIAL: NCT02604030
Title: Scapular Kinematics and Upper Limb Function in Women Who Had Undergone Breast Cancer Surgery Subjected to Upper Limb Stretching and Strengthening Exercises Program
Brief Title: Surgical Intervention and Physiotherapy in Breast Cancer: Effects in Scapular Kinematics, Pain and Upper Limb Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Ivana Leão Ribeiro, Principal Investigator, Universidade Federal de Sao Carlos
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 869.208
Record Dates: First submitted 2015-08-24; First posted 2015-11-13 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Upper limb function (Experimental): Assessment of scapular kinematics during arm elevation, perceived function, quality of life, range of motion and muscle strength for shoulder complex after a rehabilitation program focused on upper limb.
  Interventions: Other: Upper limb function

INTERVENTIONS:
Other: Upper limb function — Physical therapy program will be done in two steps, with 8 sessions each one (twice a week for four weeks). First, 8 sessions of passive mobilization in glenohumeral joint and scapular, scar massage, lymphatic drainage, stretching exercises will be completed. Second, 8 sessions of upper limb strengthening and stretching exercises for upper limb. Each session will be completed in 1 hour (twice a week) during two months.
  Other Names: Physiotherapy

SUMMARY:
Our objective is to identify the possible changes of three-dimensional scapula movement during arm elevation in women after breast cancer surgery and subjected to a physical therapy intervention. Also to evaluate pain, upper limb function and quality of life. Methods: Will be evaluated 25 women with a clinical diagnosis of breast cancer and 25 healthy controls women with no history of musculoskeletal disorders of upper limbs and matched with age and body mass index. Two pre-surgical evaluations in the month prior to surgical treatment of breast cancer and two post-surgical assessments are going to be assess: the first, after 4 weeks after surgery, when patients have received 8 sessions of physical therapy in upper limb; the second, after 8 weeks after surgery, when patients completed 16 sessions of physical therapy for shoulder complex . In each evaluation, bilateral scapular kinematics will be analyzed by an electromagnetic tracking device during arm elevation in scapula plane, in breast cancer group. Range of motion will by assessed by a digital inclinometer and muscle strength by a hand held dynamometer. Also, pain will be assessed by visual analog scale and upper limb function by DASH questionnaire. Quality of life is going to be evaluated by 36 questionnaire -item Short Form Health Survey (SF36).

DETAILED DESCRIPTION:
The main disorders of upper limb related to postoperative breast cancer, as functional limitations and muscle weakness, have already been studied. Three-dimensional scapula movement can be altered after surgical treatment of this condition, but the studies are inconclusive on this topic. Objective: To identify the possible changes of three-dimensional scapula kinematics during arm elevation in women after breast cancer surgery and subjected to a physical therapy intervention. Also to evaluate pain, upper limb function and quality of life. Methods: Will be evaluated 25 women with a clinical diagnosis of breast cancer and 25 healthy controls women with no history of musculoskeletal disorders of upper limbs and matched with age and body mass index. There will be two pre-surgical evaluations in the month prior to surgical treatment of breast cancer (with an interval of one week between then) and two post-surgical assessments: the first, after 4 weeks after surgery, when patients have received 8 sessions (twice a week) of physical therapy in upper limb (passive mobilization in glenohumeral joint and scapular, scar massage, lymphatic drainage, stretching exercises); the second, after 8 weeks after surgery, when patients completed 16 sessions (twice a week) of physical therapy for shoulder complex (strengthening and stretching exercises). In each evaluation, bilateral scapular kinematics will be analyzed by an electromagnetic tracking device during arm lifting movement in scapula plane, in breast cancer group. For control group, the assessed side will be correspondent to dominant or non-dominant operated side. Flexion, abduction, external and internal rotation of each arm will be assessed by a digital inclinometer. Muscle strength of abductors and external rotators will be evaluated by a hand held dynamometer. Pain will be assessed by visual analog scale (VAS) and upper limb function will be assessed by Disabilities of the Arm and Shoulder and Hand (DASH) questionnaire. Quality of life, through the Medical Outcomes Study 36 questionnaire -item Short Form Health Survey (SF36). Statistical analysis will include analysis of qualitative and quantitative variables. Statistical tests will be applied according to the normality of the data and it will adopt a 5% of significance level for variables comparisons along evaluations. Expected results and clinical implications of the study: To provide information of shoulder and scapular biomechanics in women after surgery for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Twenty five women with breast cancer diagnosis, more than 18 years and able to raise the arms after head level will be recruited.

Exclusion Criteria:

* History of musculoskeletal disorders of upper limbs;
* Recurrence of Breast Cancer;
* Bilateral breast cancer;
* Presence of lymphedema;
* Metastasis diagnosis;
* Attendance impact on shoulder, identified by positive tests: Hawkins - Kennedy; or shoulder injury prior to surgery, with signs and symptoms compatible with subacromial pain syndrome;
* Previous history of surgery and fractures in upper limb;
* Allergy to tape transpore, necessary to display the sensors during scapular kinematics assessment;
* Body mass index (BMI ) greater que 28 kg/m², as can compromising data quality due to increased of subcutaneous tissue amount. This has been linked to an increase in the artifact in electromagnetic kinematic analysis signal.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Three-dimensional scapular kinematics angles scores. | 1 year
  Three-dimensional scapular kinematics during arm elevation (scores are represented by movements of scapular angles at 30, 60, 90 and 120 degrees of humerus elevation).

CONTACTS AND LOCATIONS:
Locations (1):
- School healthy unity of Federal University of Sao Carlos, São Carlos, São Paulo, Brazil